CLINICAL TRIAL: NCT03088709
Title: Safety, Efficacy and Feasibility of Haploidentical Stem Cell Transplantation (Haplo-SCT) Using Post-Transplant Cyclophosphamide (PTCy) as an Alternative Donor Source for Patients Who Lack a Matched Sibling/Unrelated Donor Options
Brief Title: Haploidentical Stem Cell Transplantation Using Post-Transplant Cyclophosphamide
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Hagen, Patrick A, Assistant Professor, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 208941
Record Dates: First submitted 2017-02-22; First posted 2017-03-23 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphocytic Leukemia; Myelodysplastic Syndrome; Non-hodgkin Lymphoma; Chronic Lymphocytic Leukemia
Keywords: NHL; Non-Hodgkin Lymphoma; Haploidentical; Bone Marrow Transplant; Stem Cell Transplant; Acute Myeloid Leukemia; Acute Lymphocytic Leukemia; Myelodysplastic Syndrome; Chronic Lymphocytic Leukemia; GVHD
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All patients will receive Haploidentical (Experimental): The choice of the chemotherapy treatment for transplantation will be up to the investigator. Post-transplant cyclophosphamide will serve as the backbone of the immunosuppression treatment to prevent GVHD. All patients will receive a Haplo-identical stem cell transplantation.
  GVHD Prevention Treatment:
  Cyclophosphamide 50mg/kg will be administered IV on Day 3 and Day 5 post transplant.
  Tacrolimus 0.03 mg/kg daily will be administered IV until patient can take it by mouth starting on day of transplant and continue approximately 100 days post-transplant.
  Mycophenolate mofetil 15mg/kg will be administered twice a day IV until patient can take it by mouth starting on Day 1 post transplant until 28 days.
  Interventions: Drug: Cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Other: Haploidentical Stem Cell Transplantation

INTERVENTIONS:
Drug: Cyclophosphamide — IV medication given for prevention of graft versus host disease.
  Other Names: Cytoxan
Drug: Tacrolimus — IV medication given for prevention of graft versus host disease.
  Other Names: Prograf
Drug: Mycophenolate mofetil — IV medication given for prevention of graft versus host disease.
  Other Names: Cellcept
Other: Haploidentical Stem Cell Transplantation — A stem cell transplant that involves matching a patient's tissue type, specifically their human leukocyte antigen (HLA) tissue type, with that of a related donor.
  Other Names: Haploidentical hematopoietic stem cell transplantation

SUMMARY:
Historically, the best results of allogeneic SCT have been obtained when the stem cell donor is a human leukocyte antigen (HLA)-matched sibling, however, this is only available for approximately 30 percent of patients in need for SCT. Alternative donor sources include matched unrelated donor utilizing the donor registry, cord blood transplant and mismatched donor transplant. A human leukocyte antigen (HLA)-haploidentical donor is one who shares, by common inheritance, exactly one HLA haplotype with the recipient, and includes the biologic parents, biologic children and full or half siblings. There is strong body of evidence supporting the use of haplo-SCT in patient who lack a matched sibling or unrelated donor with high rates of successful engraftment, effective Graft Versus Host Disease (GVHD) control and favorable outcomes comparative to those seen using other allograft sources, including HLA-matched sibling SCT. Furthermore, it provides a cost-efficient donor option in a timely manner especially for patients who need to proceed quickly to transplant due to concern of disease relapse/progression.

DETAILED DESCRIPTION:
An open label, single-arm, single-center study to evaluate the safety, efficacy and feasibility of haplo-SCT as an alternative donor source for patients who lack a matched sibling/unrelated donor options. The choice of the chemotherapy treatment for transplantation will be up to the investigator. Post-transplant cyclophosphamide will serve as the backbone of the immunosuppression treatment to prevent GVHD.

GVHD Prevention Treatment:

Cyclophosphamide will be administered IV on Day 3 and Day 5 post transplant.

Tacrolimus will be administered IV until patient can take it by mouth starting on day of transplant and continue approximately 100 days post-transplant.

Mycophenolate mofetil will be administered IV until patient can take it by mouth starting on Day 1 post transplant until 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Ages 16 years old and up
* Performance Status 70 percent or above
* Patients should have the following diseases:
* Acute myelogenous leukemia (AML)
* Acute lymphocytic leukemia or lymphoblastic lymphoma (ALL)
* Transfusion dependent myelodysplastic syndrome (MDS)
* Non-Hodgkin's Lymphoma (NHL)
* Chronic lymphocytic leukemia (CLL)
* Pulmonary function as measured by forced expiratory volume at one second (FEV1) and/or corrected diffusing capacity of lung for carbon monoxide (DLCO) at 60 percent of predicted or above
* Left ventricular ejection fraction at 45 percent or above
* If the donor-specific HLA antibodies (DSA) are positive, the patient must undergo a desensitization protocol resulting in undetectable DSA prior to day of transplant

Exclusion Criteria:

* Less than twenty-one days have elapsed since the subject's last radiation or chemotherapy prior to conditioning (except for hydroxyurea)
* Uncontrolled bacterial, fungal or viral infections at time of study enrollment
* Positive for HIV, human T-cell leukemia virus (HTLV-1) and/or Hepatitis C
* Subjects with signs/symptoms of active central nervous system (CNS) disease

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Chimerism | 100 days
  Blood test that measures amount of donor's cells

SECONDARY OUTCOMES:
Neutrophil engraftment | Day 28
  Blood test that measures the white cell count
Platelet engraftment | Day 60
  Blood test that measures the platelet count
Grade 3 to 4 acute graft-verus-host disease (GVHD) | 100 days
  National Institutes of Health Acute Graft-Versus-Host Disease Grading and Form
Frequency and severity of chronic GVHD | 1 year
  National Institutes of Health Chronic Graft-Versus-Host Disease Grading and Form
Disease status with blast counts (immature blood cell count) above 5% | 3 years
  Blood work and/or bone marrow biopsy will be used
Survival status by patient contact | 3 years
  Contact with patient by phone or doctor's visit
Immune reconstitution | 3 years
  Blood work will be used to evaluate recovery of T and B cell count subset that assess cells which make antibodies to fight infections
Grade 3 through 5 Adverse Events | 2 years
  Toxicities that are possibly, probably, and definitely related to study treatment according to NCI CTCAE Version 4

CONTACTS AND LOCATIONS:
Overall Officials: Zeina Al-Mansour, MD, Principal Investigator — Cardinal Bernardin Cancer Center, Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No